CLINICAL TRIAL: NCT04903756
Title: Prediction of Risk and Communication of Outcome Following Major Lower Limb Amputation - a Collaborative Study (PERCEIVE). A Multi-methods Study of Risk Perception, Communication and the Extent and Experiences of Shared Decision Making Around the Time of Major Lower Limb Amputation.
Brief Title: The PERCEIVE Study
Acronym: PERCEIVE
Status: Completed | Type: Observational
Sponsor: Aneurin Bevan University Health Board (Other)
Collaborators: Health and Care Research Wales (Unknown)
Responsible Party: Principal Investigator, Brenig Llwyd Gwilym, Mr, Aneurin Bevan University Health Board
Other Study IDs: AB/136
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Amputation; Peripheral Artery Disease; Diabetes Mellitus
Keywords: Major lower limb amputation; Risk perception; Shared decision making
MeSH Terms: conditions — Peripheral Arterial Disease; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Adult patients where major lower limb amputation is being considered.
- Healthcare professionals: Surgeons, anaesthetists, and allied health professionals involved in decision making with patients where a major lower limb amputation is being considered.

SUMMARY:
The PERCEIVE (PrEdiction of Risk and Communication of outcomE followIng major lower limb amputation - a collaboratiVE study) study aims to explore how decisions about major lower limb amputations are made by patients and healthcare professionals.

DETAILED DESCRIPTION:
This study will look in detail at major lower limb amputation risk perception, communication and decision-making, both from a patient/family and a surgeon/clinician point of view. The investigators will audio-record 10-15 consultations between surgeons and patients, examining the communication and decision-making process, and conduct individual interviews with 10-15 patients and 10-15 healthcare professionals. Patients will be interviewed at two time points: firstly as soon as possible after they discuss the possibility of leg amputation with a surgeon, and secondly around six months later. The investigators will identify what is important to patients, what information they need to make an informed decision and how best to communicate that information. Interviews with surgeons, anaesthetists and specialist physiotherapists will explore how they estimate risks and outcomes of amputation surgery, and how they communicate this to patients. Finally, the investigators will combine all this information together and discuss our findings with groups of patients and healthcare professionals, to identify key areas around amputation decision-making that can be improved and how best to further examine those areas.

ELIGIBILITY:
Inclusion Criteria:

* Any patient aged 18 years old or over with chronic limb threatening ischaemia or diabetic foot disease for whom major lower limb amputation is considered or discussed
* Vascular surgeons / anaesthetists / specialist physiotherapists involved in, or supporting major lower limb amputation decision making

Exclusion Criteria:

* Patients under 18 years old
* Patients undergoing major lower limb amputation for other causes (e.g. trauma or cancer)
* Any patient/healthcare professional unable or unwilling to provide informed consent. Some patients undergoing emergency major lower limb amputation will have insufficient time to give informed consent
* Potential participants with an insufficient understanding of English or Welsh to be able to provide informed consent
* Potential participants unable to complete an interview in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are eligible for the study if they meet all of the following inclusion criteria and none of the exclusion criteria apply. All queries about participant eligibility should be directed to the Qualitative Researcher. We will purposively sample participants from up to four participating NHS Health Boards / Trusts in Wales and England. We will aim to include 8-10 surgeons, 1-3 anaesthetists and 1-3 specialist physiotherapists from several Health Boards / Trusts. We will purposively sample patients for inclusion in the audio-recorded consultations and interviews to ensure our sample has variation in terms of gender, age, MLLA type (above knee/below knee/no amputation) and Health Board / Trust.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Analysis of audio-recorded consultations between surgeons and patients. | During primary consultation
  Theme-oriented discourse analysis

SECONDARY OUTCOMES:
Analysis of patient interviews | As soon as possible after the time of consultation and approximately 6 months following consultation
  Thematic analysis of interview transcripts
Analysis of healthcare professional interviews | As soon as possible after the time of consultation
  Thematic analysis of interview transcripts

CONTACTS AND LOCATIONS:
Locations (1):
- Aneurin Bevan University Health Board, Newport, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Prout H, Waldron CA, Gwilym B, Thomas-Jones E, Milosevic S, Pallmann P, Harris D, Edwards A, Twine CP, Massey I, Burton J, Stewart P, Jones S, Cox D, Bosanquet DC, Brookes-Howell L; PERCEIVE Study group; PERCEIVE Study. Challenges in shared decision-making about major lower limb amputation: the PERCEIVE qualitative study. BMJ Open. 2026 Jan 12;16(1):e104407. doi: 10.1136/bmjopen-2025-104407. PMID 41526012